CLINICAL TRIAL: NCT06391411
Title: : Effect of Supplementation With Lutein, Zeaxanthin and Saffron on the Intestinal Microbiota in Patients Suffering From Age-related Macular Degeneration - The Gut-Retina-axis Study"
Brief Title: Effect of Micronutrient Supplementation on the Intestinal Microbiota in Patients With Age-related Macular Degeneration - The Gut-Retina-axis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: Azienda USL Toscana Centro (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Associate Professor of Clinical Nutrition, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Drusen off
Record Dates: First submitted 2024-04-16; First posted 2024-04-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; Gut microbiota; Gut-retina axis; Micronutrient; Short chain fatty acids
MeSH Terms: conditions — Macular Degeneration | interventions — Zeaxanthins; Ascorbic Acid; Vitamin E; Zinc

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Healthy controls received no intervention
- Micronutrient supplementation+ Aflibercept 2 mg, 0.05 ml (Experimental): Patients received intravitreal injections of anti-VEGF (Aflibercept 2 mg, 0.05 ml) at a fixed regimen and daily supplementation with a micronutrient mix containing lutein (10 mg), zeaxanthin (2 mg), saffron (20 mg), vitamin C (80 mg), vitamin E (12 mg) and zinc (10mg) for 6 months
  Interventions: Dietary Supplement: a micronutrient mix containing lutein (10 mg), zeaxanthin (2 mg), saffron (20 mg), vitamin C (80 mg), vitamin E (12 mg) and zinc (10mg); Drug: anti-VEGF treatment
- Aflibercept 2 mg, 0.05 ml (Active Comparator): Patients received only intravitreal injections of anti-VEGF (Aflibercept 2 mg, 0.05 ml) for 6 months
  Interventions: Drug: anti-VEGF treatment

INTERVENTIONS:
Dietary Supplement: a micronutrient mix containing lutein (10 mg), zeaxanthin (2 mg), saffron (20 mg), vitamin C (80 mg), vitamin E (12 mg) and zinc (10mg) — In this three-arm randomized, controlled trial, with one arm represented by healthy subjects, eligible participants were randomly divided into two groups. Fifteen patients were randomly allocated to the intervention group and received, for 6 months, intravitreal injections of anti-VEGF (Aflibercept 2 mg, 0.05 ml) at a fixed regimen and daily supplementation with a micronutrient mix containing lutein (10 mg), zeaxanthin (2 mg), saffron (20 mg), vitamin C (80 mg), vitamin E (12 mg) and zinc (10mg). The other fifteen patients was assigned to the control group and only received the intravitreal anti-VEGF treatment at a fixed regimen for 6 months
  Other Names: Drusen off
  Arms: Micronutrient supplementation+ Aflibercept 2 mg, 0.05 ml
Drug: anti-VEGF treatment — Intravitreal injections of anti-VEGF (Aflibercept 2 mg, 0.05 ml) at a fixed regimen for six months
  Arms: Aflibercept 2 mg, 0.05 ml; Micronutrient supplementation+ Aflibercept 2 mg, 0.05 ml

SUMMARY:
Age-related macular degeneration (AMD) is a leading cause of visual impairment in the elderly, characterized by multifactorial etiology. Recent evidence suggests a potential involvement of the gut-retina axis in AMD pathogenesis, prompting exploration into novel therapeutic strategies. The investigators assessed the effects of a micronutrient mix containing lutein, zeaxanthin, and saffron, recognized for their anti-inflammatory properties, on ophthalmological and microbial parameters in neovascular AMD (nAMD) patients. Thirty nAMD subjects were randomized to receive daily micronutrient supplementation along with anti-VEGF therapy or anti-VEGF treatment alone for 6 months. Ophthalmological assessments, anthropometric and biochemical measurements and stool samples were obtained pre- and post-treatment. Gut microbiota (GM) characterization was performed through 16S rRNA sequencing while short (SCFAs), medium (MCFAs) and long (LCFAs) chain fatty acids were analyzed with a gas chromatography-mass spectrometry protocol. nAMD patients exhibited reduced GM alpha diversity, altered taxonomic abundances and decreased total SCFA amount, coupled with elevated proinflammatory octanoic and nonanoic acids. Micronutrient supplementation led to improved visual acuity in comparison to the control group, along with the reduction in the total amount of MCFAs, metabolites exerting detrimental ocular effects. This study reveals compositional and functional imbalances in the GM of nAMD patients compared to healthy controls. Furthermore micronutrient supplementation demonstrated a potential to restore the gut-retina axis, suggesting its therapeutic efficacy in improving ocular outcomes in nAMD patients. These findings underscore the intricate interplay between the GM and ocular health, offering insights into innovative interventions for AMD management

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) stands as the primary cause of visual impairment in the over-65-year-old population of industrialized countries, affecting approximately 170 million people worldwide . AMD is a multifactorial disease in the pathogenesis of which, that it's not yet fully understood, genetic and environmental factors are involved. Specifically, there are two main types of AMD, both culminating in central vision deficiency and potential blindness due to the death of photoreceptors. The first type of AMD type, known as dry AMD, is characterized by the accumulation of extracellular material (i.e. lipids, vitronectin, inflammatory or amyloid proteins) between the Bruch's membrane and the retinal pigment epithelium, leading to the formation of drusen. Drusen are small yellow or white spots on the retina that can gradually evolve either into retinal and pigment epithelium atrophy or, for approximately 20% of patients, progress into the second AMD type that is called wet AMD or neovascular AMD (nAMD). nAMD is distinguished by the development of new choroidal vessels, a condition that can result in permanent visual impairment. Presently, although therapeutic options for dry AMD are limited, nAMD is treated with intravitreal injections of anti-VEGF (vascular endothelial growth factor) drugs, which have proven effective in slowing angiogenic development and limiting the progression of nAMD. Moreover, recent investigations have implicated immune system alterations, oxidative stress, and overweight as critical factors in AMD pathogenesis. Particularly, many studies have recently highlighted the potential benefits of dietary supplementation with micronutrients having antioxidant and antiinflammatory effects in reducing the risk of AMD development. Notably, the AREDS2 study definitively demonstrated the efficacy of dietary supplementation with lutein and zeaxanthin in reducing the risk of progression of early-stage AMD. In detail, the administration of lutein and zeaxanthin, which can absorb blue light and neutralize free radicals and reactive oxygen species in the macula, has been associated with increased macular pigment optical density (MPOD), improved visual acuity and a reduced risk of retinal aging. Moreover, other micronutrients such as vitamins E and C can prevent the progression of maculopathy by providing protection against oxidative stress and maintaining GM homeostasis while oral zinc supplementation can reduce the complement-mediated inflammation in the retinal pigment epithelium, which plays a fundamental role in the etiology of AMD. Additionally, saffron (Crocus sativus), which contains active components such as crocin, safranal, crocetin, and picrocrocin, has demonstrated antioxidant and anti-inflammatory effects, leading to significant improvements in the retinal function of AMD patients. Furthermore, considering that the retina is an extension of the brain both anatomically and developmentally, the hypothesis of a gut-retina interplay has been recently proposed, paralleling the widely explored bidirectional communication between the gut and the brain. Objectives of the study To evaluate the GM composition and function of nAMD patients in comparison to healthy subjects and considering the dual potential of micronutrients to act through direct antioxidant mechanisms and modulation of the GM, the investigators assessed the impact of a novel micronutrient supplementation based on lutein, zeaxanthin and saffron on ophthalmological parameters and microbial features of nAMD patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >50 years of age.
* Willingness to cooperate during the study and ability to follow guidelines and to complete all clinical visits
* Ability to provide informed consent

Exclusion Criteria:

* Use of antibiotics or continued use of pre- or probiotics in the 2 months before enrolment
* Use of other treatments (medications or nutritional programs) that affect body weight, food intake, and/or energy expenditure
* Diagnosis of any ocular disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota composition | At baseline and at month 6
  Changes in gut microbiota composition assessed by 16S sequencing
Changes in gut microbiota function | At baseline and at month 6
  Changes in gut microbiota function (quantification of short-, medium- and long-chain fatty acids)assessed with gas chromatography-mass spectrometry
Ophthalmological examination | At baseline and at month 6
  Ophthalmological examination with best correct visual acuity (BCVA), biomicroscopy and swept optical coherence tomography (OCT)

SECONDARY OUTCOMES:
White blood cells | At baseline and at month 6
  Quantification with standard laboratory procedures
Red blood cells | At baseline and at month 6
  Quantification with standard laboratory procedures
Hemoglobin | At baseline and at month 6
  Quantification with standard laboratory procedures
Platelets | At baseline and at month 6
  Quantification with standard laboratory procedures
Glucose | At baseline and at month 6
  Quantification with standard laboratory procedures
HDL-cholesterol | At baseline and at month 6
  Quantification with standard laboratory procedures
LDL-cholesterol | At baseline and at month 6
  Quantification with standard laboratory procedures
Triglycerides | At baseline and at month 6
  Quantification with standard laboratory procedures
Evaluation of Interleukin-6 | At baseline and at month 6
Evaluation of Interleukin-10 | At baseline and at month 6
Evaluation of tumor necrosis factor-α (TNF-α) | At baseline and at month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pennington KL, DeAngelis MM. Epidemiology of age-related macular degeneration (AMD): associations with cardiovascular disease phenotypes and lipid factors. Eye Vis (Lond). 2016 Dec 22;3:34. doi: 10.1186/s40662-016-0063-5. eCollection 2016. PMID 28032115
- [Result] Rein DB, Wittenborn JS, Zhang X, Honeycutt AA, Lesesne SB, Saaddine J; Vision Health Cost-Effectiveness Study Group. Forecasting age-related macular degeneration through the year 2050: the potential impact of new treatments. Arch Ophthalmol. 2009 Apr;127(4):533-40. doi: 10.1001/archophthalmol.2009.58. PMID 19365036
- [Result] Chapman NA, Jacobs RJ, Braakhuis AJ. Role of diet and food intake in age-related macular degeneration: a systematic review. Clin Exp Ophthalmol. 2019 Jan;47(1):106-127. doi: 10.1111/ceo.13343. Epub 2018 Jul 10. PMID 29927057
- [Result] Rinninella E, Mele MC, Merendino N, Cintoni M, Anselmi G, Caporossi A, Gasbarrini A, Minnella AM. The Role of Diet, Micronutrients and the Gut Microbiota in Age-Related Macular Degeneration: New Perspectives from the Gut(-)Retina Axis. Nutrients. 2018 Nov 5;10(11):1677. doi: 10.3390/nu10111677. PMID 30400586
- [Result] Zhang QY, Tie LJ, Wu SS, Lv PL, Huang HW, Wang WQ, Wang H, Ma L. Overweight, Obesity, and Risk of Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2016 Mar;57(3):1276-83. doi: 10.1167/iovs.15-18637. PMID 26990164
- [Result] Age-Related Eye Disease Study 2 (AREDS2) Research Group; Chew EY, Clemons TE, Sangiovanni JP, Danis RP, Ferris FL 3rd, Elman MJ, Antoszyk AN, Ruby AJ, Orth D, Bressler SB, Fish GE, Hubbard GB, Klein ML, Chandra SR, Blodi BA, Domalpally A, Friberg T, Wong WT, Rosenfeld PJ, Agron E, Toth CA, Bernstein PS, Sperduto RD. Secondary analyses of the effects of lutein/zeaxanthin on age-related macular degeneration progression: AREDS2 report No. 3. JAMA Ophthalmol. 2014 Feb;132(2):142-9. doi: 10.1001/jamaophthalmol.2013.7376. PMID 24310343
- [Result] Zeng S, Hernandez J, Mullins RF. Effects of antioxidant components of AREDS vitamins and zinc ions on endothelial cell activation: implications for macular degeneration. Invest Ophthalmol Vis Sci. 2012 Feb 27;53(2):1041-7. doi: 10.1167/iovs.11-8531. Print 2012 Feb. PMID 22247465